CLINICAL TRIAL: NCT00261560
Title: A Randomized, Double-Blind, Parallel-Group Study Comparing the Safety and Effectiveness of Acetaminophen Extended Release (3900 mg/Day) and Ibuprofen (1200 mg/Day) in the Treatment of Ankle Sprains.
Brief Title: A Safety and Effectiveness Study of Acetaminophen Extended Release (3900 mg/Day) and Ibuprofen (1200 mg/Day) in the Treatment of Pain Associated With Ankle Sprains.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002824
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Sprains and Strains; Pain
Keywords: ankle sprain; acetaminophen extended release, ibuprofen
MeSH Terms: conditions — Sprains and Strains; Pain; Ankle Injuries | interventions — Acetaminophen

INTERVENTIONS:
Drug: acetaminophen

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of 1300 mg acetaminophen extended release given three times daily for nine days to that of 400 mg ibuprofen given three times daily for nine days for the signs and symptoms of (Grade I and Grade II) lateral ankle sprains.

DETAILED DESCRIPTION:
The objective of this randomized, double-blind, parallel-group study is to compare the safety and effectiveness of 1300 mg acetaminophen extended release given three times daily for nine days to that of 400 mg ibuprofen given three times daily for nine days for the signs and symptoms of Grade I and Grade II lateral ankle sprains. The primary efficacy endpoint is the change from baseline (Day 1) to Day 4 in the subjects' pain upon walking. Safety assessments consist of the monitoring of adverse events and assessments of the ankle injury during the course of the study. Two hypotheses are examined using a step down approach. The first hypothesis is that acetaminophen extended release is not inferior to ibuprofen in relieving the pain associated with (Grade I or Grade II) lateral ankle sprains. If acetaminophen extended release is not inferior to ibuprofen in relieving the pain associated with Grade I or Grade II lateral ankle sprains, the second hypothesis is that acetaminophen extended release is superior to ibuprofen in relieving the pain associated with Grade I or Grade II lateral ankle sprains. Two acetaminophen 650 mg extended release caplets, taken by mouth, three times a day for nine days or two ibuprofen 200 mg caplets, taken by mouth, three times a day for nine days

ELIGIBILITY:
Inclusion Criteria:

* Have had an ankle sprain within 24 hours of study entry
* have ankle pain when walking
* have not recently used non-steroidal, anti-inflammatory drugs (NSAIDs), other pain relieving medications (including acetaminophen) or medicines that could interfere with the assessment of effectiveness
* if female, must not be pregnant or breastfeeding

Exclusion Criteria:

* Ankle sprain was the second ankle sprain within six months
* Both ankles were sprained
* Ankle sprain occurred on the same side of the body as a knee injury
* Ankle injury requires bed rest, hospitalization, surgical intervention, or use of a non-removable rigid cylindrical cast
* Subject reports severe or very severe pain at rest on a five-point scale of none, mild, moderate, severe or very severe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Day 1) to Day 4 in the subject's pain upon walking using a 0 to 100 mm visual analogue scale.

SECONDARY OUTCOMES:
Change from baseline to Day 9 in pain upon walking; change from baseline to Day 4 and 9 in: ability to walk, ankle swelling, ankle bruising, and ankle's range of motion; overall satisfaction with treatment from Day 1 to Day 4 and Day 1 to Day 9.

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Result] Dalton JD Jr, Schweinle JE. Randomized controlled noninferiority trial to compare extended release acetaminophen and ibuprofen for the treatment of ankle sprains. Ann Emerg Med. 2006 Nov;48(5):615-23. doi: 10.1016/j.annemergmed.2006.05.015. Epub 2006 Sep 1. PMID 17052565